CLINICAL TRIAL: NCT02517502
Title: Docosahexaenoic Acid (DHA) To Prevent Development of Cognitive Dysfunction Due to Chemotherapy
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: Carol Fabian, MD (Other)
Collaborators: DSM Nutritional Products, Inc. (Industry)
Responsible Party: Sponsor-Investigator, Carol Fabian, MD, Professor, Director Breast Cancer Prevention Unit, University of Kansas Medical Center
Organization: University of Kansas Medical Center (Other)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Supportive Care
Other Study IDs: STUDY00002415
Record Dates: First submitted 2015-07-08; First posted 2015-08-07 (Estimated); Last update posted 2022-01-24 (Actual); Status verified 2021-03

CONDITIONS: Cognitive Dysfunction
Keywords: DHA; Omega-3; neoadjuvant chemotherapy; chemotherapy; breast cancer
MeSH Terms: conditions — Cognitive Dysfunction; Breast Neoplasms | interventions — Docosahexaenoic Acids

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- DHA (Experimental): Participants will be asked to take four 400 mg (1600 mg; 1.6 grams) capsules of DHA daily. Participants will start taking capsules before the start of and for the duration of their neoadjuvant chemotherapy.
  Interventions: Drug: DHA
- Placebo (Placebo Comparator): Participants will be asked to take four 400 mg (1600 mg; 1.6 grams) capsules of a matched placebo daily. Participants will start taking capsules before the start of and for the duration of their neoadjuvant chemotherapy.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: DHA — 4 capsules of 400 mg DHA daily
  Other Names: Docosahexaenoic Acid
  Arms: DHA
Drug: Placebo — Matched, blinded placebo
  Arms: Placebo

SUMMARY:
The purpose of this study is to determine if a high dose of DHA begun prior to and continued during neo-adjuvant chemotherapy (chemotherapy given prior to surgery) is likely to prevent or lessen chemotherapy induced cognitive dysfunction.

DETAILED DESCRIPTION:
Chemotherapy is often associated with problems of cognitive functioning such as decision making, learning, and memory. These symptoms, collectively referred to here as cognitive dysfunction can appear as early as the first few months after starting chemotherapy and may persist long after chemotherapy and anti-hormone therapy, if any, is completed.

Once developed there is no satisfactory treatment for cognitive dysfunction although cognitive retraining and exercise may improve symptoms and/or function; at least for some.

Omega-3 fatty acids derived from ocean fish are a new potential preventative treatment against development of cognitive problems which can arise in some individuals during chemotherapy treatment. In doses of 1-2 grams per day it has been found to improve some aspects of cognitive function in healthy adults who have low DHA dietary intake. It has also been shown to improve some aspects of function in individuals with a mild reduction in cognitive ability but not for those with marked impairment.

Participation in this study will last about 12 months. Participants will make visits to the study site for both standard of care visits and additional study-related visits. Participants will be randomized (randomly assigned; like flipping a coin) to one of two groups. Neither the Investigator nor the participant will know the assigned treatment.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of invasive breast cancer (Stage I-III) and are anticipated to start neo-adjuvant chemotherapy (multiple chemotherapy regimens allowed under protocol)
* Able to read, write, and understand English and at least have a high school education.
* Able and willing to go at least 24-36 hours without narcotic pain medicine, muscle relaxants, sedatives, sleeping pills and alcohol prior to their cognitive testing. Participants should not have required chronic sedatives, sleeping aids, or narcotic pain medications on a daily basis prior to their diagnosis.
* Willing to complete required study procedures from start of study to approximately 6 months after completion of neo-adjuvant chemotherapy.

Exclusion Criteria:

* Women who are currently on omega-3 fatty acid supplements with > 500 mg of EPA plus DHA daily or 250 mg of DHA alone and or who have chronically been on more than 1 fish oil capsule per day.
* Individuals who are not willing to stop fish or krill oil supplements during the study.
* Diabetics requiring insulin treatment.
* Individuals who are not likely to be able to go for 24 hours without sleeping pills, sedatives, narcotic pain medications, or ativan
* Individuals who do not have a high school education or are not fluent in English.
* Individuals who have already started chemotherapy for breast cancer or who have previously had systemic chemotherapy for a malignancy.
* Women who have already had definitive surgery for breast cancer.

Ages: 18 Years to 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2015-07; Primary Completion 2017-09 (Actual); Study Completion 2019-05-03 (Actual)

PRIMARY OUTCOMES:
Trial acceptance | 12 months
  Number of potentially eligible subjects who consent to participate in the study.
Subject retention and trial completion | Completion of study (~12 months)
  Number of enrolled subjects who complete all cognitive assessments at all three defined timepoints.
Compliance with taking study agent. | Completion of study (~12 months)
  Number of enrolled subjects who take at least 70% of prescribed study agent.
Number of subjects reporting serious adverse events | Completion of study (~12 months)
  Number of enrolled subjects randomized to DHA who report serious adverse events (adjusted for subjects randomized to placebo who report serious adverse events).

SECONDARY OUTCOMES:
Change in Cognitive Ability-General Concerns Questionnaire | Baseline to Month 12
  Change measured using Patient-Reported Outcomes Measurement Information System (PROMIS-General Concerns). There are a total of 34 questions. Each question has five response options ranging in value from one to five (never to very often). The total score is based on the sum of the responses, multiplied by the number of questions and then divided by the number of questions that were answered.
Change in Cognitive Ability-Abilities Questionnaire | Baseline to Month 12
  Change measured using Patient-Reported Outcomes Measurement Information System (PROMIS-Abilities). There are a total of 33 questions. Each question has five response options ranging in value from one to five (never to very often). The total score is based on the sum of the responses, multiplied by the number of questions and then divided by the number of questions that were answered.
Change in Quality of Life Questionnaire | Baseline to Month 12
  Change measured using Patient-Reported Outcomes Measurement Information System (PROMIS 29-Profile). The PROMIS 29-Profile includes 4 items from 7 different domains (Depression, Anxiety, Physical Function, Pain Interference, Fatigue, Sleep Disturbance, and Ability to Participate in Social Roles and Activities, along with a single item on pain intensity). The total score is based on the sum of the responses, multiplied by the number of questions and then divided by the number of questions that were answered.
Level of Physical Activity Questionnaire | Month 12
  Physical activity will be tracked over course of the study. Participants will complete a physical activity questionnaire (PAQ-4) at each visit.
Change in Cognitive Function test | Change from Baseline to Month 12
  Change measured based on standard battery of cognitive tests including Hopkins Verbal Learning Test-Revised, Trail Making A, Trail Making B and Controlled Oral Word Association.
Measurement of Cognitive Function Mobile Cognitive Assessment Battery (MCAB) Questionnaire | Change from Baseline to Month 12
  The MCAB measures working memory, divided attention/multitasking, cognitive flexibility and processing speed and also includes a 33 item self-rating questionnaire that assesses everyday cognitive behaviors, physical activity, sleep, pain and functional adjustment.

CONTACTS AND LOCATIONS:
Overall Officials: Carol Fabian, MD, Principal Investigator — University of Kansas Medical Center
Locations (2):
- United States (2):
  - Decatur Memorial Hospital, Decatur, Illinois
  - University of Kansas Medical Center, Kansas City, Kansas

IPD SHARING:
Plan to Share IPD: No
Global results will be published.